CLINICAL TRIAL: NCT06101628
Title: Effect of Gel Nail Application on Pulse Oximetry Measurements in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other); Necmettin Erbakan University (Other); Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Research Assistant, Tarsus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TU-BOZKUL-004
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy Individuals; Gel Nail; Oxygen Saturation; Nursing; Perioperative Care

STUDY DESIGN:
Intervention Model Description: This study is a prospective, self-controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXPERIMENTAL AND CONTROL GROUP (Other): Participants who meet the inclusion criteria of the study will be informed about the research by the researchers and will be included in the study on a voluntary basis and their written permissions will be obtained. Firstly, the personal information of the participants will be recorded in the data collection form. The middle finger of the left hand of each participant will be the experimental group and the little finger will be the control group. After the gel nail is applied to the middle finger of the left hand, SpO2 and pulse values will be measured by pulse oximetry from the left hand middle finger and little finger of the participant and recorded in the data form. At the end of the study, SpO2 and pulse values before and after the gel nail application will be compared.
  Interventions: Other: Gel nail application

INTERVENTIONS:
Other: Gel nail application — The middle finger of the left hand of each participant will be the experimental group and the little finger will be the control group. After the gel nail is applied to the middle finger of the left hand, SpO2 and pulse values will be measured by pulse oximetry from the left hand middle finger and little finger of the participant
  Other Names: Control group: Non-applied nail

SUMMARY:
The aim of this study was to determine the effect of gel nail application on pulse oximetry measurements in healthy subjects. This study was planned as a prospective, self-controlled clinical research to determine the effect of gel nail application on SpO2 and pulse values in healthy people. The population of the study will consist of women who had gel nail application in a private beauty centre between July 2023 and October 2023. The minimum required sample size was calculated as 162 in G*Power (3.1.9.2) programme (α=0.05 (two-way), 1-β=0.95). The data will be collected with the data collection form prepared in line with the literature. Firstly, the personal information of the participants will be recorded in the data collection form. The middle finger of the left hand of each participant will be the treatment group and the little finger will be the control group. After the gel nail is applied to the middle finger of the left hand, SpO2 and pulse values will be measured simultaneously with a pulse oximeter from the left hand middle finger and little finger of the participant and recorded on the data form. The data obtained from the study will be analysed using SPSS (Statistical Package for Social Sciences) for Windows 26.0 software.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of gel nail application on pulse oximetry measurements in healthy subjects. This study was planned as a prospective, self-controlled clinical research to determine the effect of gel nail application on SpO2 and pulse values in healthy people. The population of the study will consist of women who had gel nail application in a private beauty centre between July 2023 and October 2023. The minimum required sample size was calculated as 162 in G*Power (3.1.9.2) programme (α=0.05 (two-way), 1-β=0.95). The data will be collected with the data collection form prepared in line with the literature.On this form, the age of the individual, the color of the gel nail, smoking status, and the SpO2 and pulse values measured by pulse oximetry from the little and middle finger will be recorded. SpO2 and pulse rates will be measured with a calibrated Jumper pulse oximeter. Since the gel nail and non-gel nail will be measured at the same time, two of the same brand pulse oximeter devices will be provided.Volunteers who meet the inclusion criteria of the research will be informed about the research and will be included in the research on a voluntary basis and their written consent will be obtained. Firstly, the personal information of the participants will be recorded in the data collection form. The middle finger of the left hand of each participant will be the treatment group and the little finger will be the control group. After the gel nail is applied to the middle finger of the left hand, SpO2 and pulse values will be measured simultaneously with a pulse oximeter from the left hand middle finger and little finger of the participant and recorded on the data form. The data obtained from the study will be analysed using SPSS (Statistical Package for Social Sciences) for Windows 26.0 software. Mean and standard deviation will be used in the evaluation of the data. Statistical significance will be accepted as p<0.05 (95% confidence interval).

ELIGIBILITY:
Inclusion Criteria:

* No communication problems,
* With full left-hand fingernails,
* No structural problems such as clubbing,
* Body temperature ≥ 36- <37.5 ºc,
* SpO2 value ≥ 95%,
* Capillary refill ≤ 2 seconds,
* Who volunteered to participate in the research,
* No psychiatric or physical illness that prevents communication,
* Without circulatory problems such as Reynauld syndrome and peripheral arterial disease,
* Without anaemia,
* No respiratory diseases such as chronic obstructive pulmonary disease and asthma
* Becoming a woman

Exclusion Criteria:

* Communication problems,
* Incomplete left fingernails,
* Structural problems like sticky fingers,
* Body temperature ≥ 36- < 37.5 ºc,
* SpO2 value <95%,
* Capillary refill >2 seconds,
* Not volunteering to participate in the research,
* Psychiatric or physical illness that prevents communication,
* With circulatory problems such as Reynauld syndrome and peripheral arterial disease,
* Anaemia
* Respiratory diseases such as chronic obstructive pulmonary disease and asthma
* Not being of the female gender

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
SpO2 value | 3 months
  Data collection form: After the gel nail was applied to the middle finger of the left hand, SpO2 values were measured and recorded by pulse oximetry from the left hand middle finger and little finger of the participant.
Pulse value | 3 months
  Data collection form: After the gel nail was applied to the middle finger of the left hand, pulse values were measured and recorded by pulse oximetry from the left hand middle finger and little finger of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, Assoc. Dr., Principal Investigator — Mersin University; Ayşenur Serbest Baz, Lecturer, Principal Investigator — Mustafa Kemal University; Serpil Yüksel, Assoc.Dr., Principal Investigator — Necmettin Erbakan University
Locations (1):
- Gamze Bozkul, Mersin, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aggarwal AN, Agarwal R, Dhooria S, Prasad KT, Sehgal IS, Muthu V. Impact of Fingernail Polish on Pulse Oximetry Measurements: A Systematic Review. Respir Care. 2023 Sep;68(9):1271-1280. doi: 10.4187/respcare.10399. Epub 2023 Apr 25. PMID 37185113
- [Background] Ballesteros-Pena S, Fernandez-Aedo I, Picon A, Lorrio-Palomino S. [Influence of nail polish on pulse oximeter readings of oxygen saturation: a systematic review]. Emergencias. 2015 Oct;27(5):325-331. Spanish. PMID 29087059
- [Background] Cabanas AM, Fuentes-Guajardo M, Latorre K, Leon D, Martin-Escudero P. Skin Pigmentation Influence on Pulse Oximetry Accuracy: A Systematic Review and Bibliometric Analysis. Sensors (Basel). 2022 Apr 29;22(9):3402. doi: 10.3390/s22093402. PMID 35591092
- [Background] Deniz Dogan S, Karacay Yikar S, Arslan S, Nazik E. The Effect of Nail Polish and Henna on the Measures of Pulse Oximeters in Healthy Persons. J Perianesth Nurs. 2021 Oct;36(5):532-535. doi: 10.1016/j.jopan.2020.10.013. Epub 2021 Apr 26. PMID 33926803
- [Background] Desalu I, Diakparomre OI, Salami AO, Abiola AO. The effect of nail polish and acrylic nails on pulse oximetry reading using the Lifebox oximeter in Nigeria. Niger Postgrad Med J. 2013 Dec;20(4):331-5. PMID 24633278
- [Background] Hafen BB, Sharma S. Oxygen Saturation. (2022). In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2023 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK525974/